CLINICAL TRIAL: NCT04031235
Title: A Randomized Controlled Trial Comparing a Children's Book to Brochures for Safe Sleep and Infant Reading Education During Prenatal Obstetric Visits
Brief Title: Comparing Children's Books to Brochures for Safe Sleep and Infant Reading Education During Prenatal Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: University of Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2018-5564
Record Dates: First submitted 2019-02-16; First posted 2019-07-24 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Sudden Unexplained Infant Death; Child Rearing; Literacy
MeSH Terms: conditions — Literacy

STUDY DESIGN:
Who Masked: Participant
Masking Description: Mothers will be blinded as to the specific aims of the study other than that it involves "safe sleep and reading with your baby."
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Safe Sleep Education (Experimental): Mothers in the intervention group will receive education on American Academy of Pediatrics safe sleep recommendations using a specially-designed children's book (Sleep Baby, Safe and Snug). In addition, they will receive information on the importance of reading with their infant using a brochure created by the AAP.
  Interventions: Behavioral: Sleep Baby, Safe and Snug
- Infant Reading Education (Active Comparator): Mothers in the control group will receive education on American Academy of Pediatrics recommendations on reading and talking to infants using a specially-designed children's book (Read Baby, Every Day). In addition, they will receive information on safe sleep using a brochure created by the AAP.
  Interventions: Behavioral: Read Baby, Every Day

INTERVENTIONS:
Behavioral: Sleep Baby, Safe and Snug — Specially designed children's book, 14 pages, rhyming, illustrated in color, written at a Kindergarten reading level. Each page spread highlights AAP-recommended safe sleep practices. AAP safe sleep recommendations listed on the back cover.
  Arms: Safe Sleep Education
Behavioral: Read Baby, Every Day — Specially designed children's book, 14 pages, rhyming, illustrated in color, written at a Kindergarten reading level. Each page spread highlights AAP-recommendations regarding the importance of reading and talking to infants. Recommendations and benefits of reading with infants are listed on the back cover as well.
  Arms: Infant Reading Education

SUMMARY:
The aim of this randomized trial is to compare a specially designed children's book to brochures for safe sleep education via clinical providers at a third trimester prenatal obstetric visit. Mothers in the control group will receive a specially designed children's book regarding the importance of reading with their infant at this visit, compared to brochures. Knowledge of safe sleep and home literacy orientation will be assessed at baseline prenatally, and their first postpartum obstetric visit.

DETAILED DESCRIPTION:
This study is a randomized controlled trial (RCT) involving 2 groups of pregnant women from low-socioeconomic status (SES) backgrounds at-risk for adverse cognitive and health outcomes for their infant. Mothers will be randomly assigned to intervention and control groups during a third-trimester prenatal visit at a hospital-affiliated obstetric clinic, via convenience sampling. Mothers in the intervention group will receive education on American Academy of Pediatrics (AAP) safe sleep recommendations using a specially-designed children's book (Sleep Baby, Safe and Snug), while those in the control group will receive this guidance via a brochure endorsed by the AAP.

In a "mirror" design, mothers in the control group will receive guidance on reading with their infant using a specially designed children's book (Read Baby, Every Day), and mothers in the intervention group will receive guidance on reading with their infant using a brochure created and endorsed by the AAP.

Clinical research coordinators (CRCs) will obtain consent and collect data at two time points: 1) a 3rd trimester prenatal visit (approximately 36-38 weeks estimated gestational age; baseline), and 2) at the first, regularly scheduled postpartum visit (4-6 weeks after delivery for an uncomplicated vaginal delivery, and 2 weeks for cesarean section). Data will be collected in 4 categories, which will be compared between groups: 1) demographics, 2) maternal knowledge of AAP safe sleep recommendations, 3) maternal attitudes about reading with infants, 4) maternal impression of the printed educational materials provided, and 4) clinician impression of the feasibility and usefulness of the printed materials provided for obstetric prenatal care.

Educational materials will be shared with mothers by obstetric providers (obstetric attending physicians and residents) during this visit, who will be provided with a brief summary of content and to conduct the visit as they see fit. Mothers will be blinded to the aims of the study, other than that it is to "share information about safe sleep and reading with your baby."

ELIGIBILITY:
Inclusion Criteria:

1. confirmed viable pregnancy, with estimated gestational age (EGA) of at least 36 weeks at the baseline/enrollment prenatal visit,
2. maternal age at least 16 years old,
3. comfort speaking English during their visit and reviewing/comprehending study materials without a translator.

Exclusion Criteria:

Non-meeting the above.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant mothers
Enrollment: 144 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Safe Sleep Knowledge | Baseline prenatal (>= 32 weeks) and postpartum (<= 6 weeks).
  The safe sleep assessment is based on a version developed by the PI and used in a recent published study, reflecting current AAP guidelines. Three questions are adapted from a published survey, gauging the mother's familiarity with SUID/SIDS (and briefly explaining if unfamiliar), whether she personally knows anyone who has lost a child to SUID/SIDS, and level of worry about SUID/SIDS for her baby. Our primary knowledge question utilizes an open-ended format, as no established tool for measuring SIDS knowledge was available: "Name as many things as you can think of to help keep your baby safe from SUID/SIDS (dying while asleep)." Maternal responses will be compared to an 11-item checklist of AAP safe sleep recommendations which are each referenced at least once in the book and brochures used, with 1 point awarded for each correct response.
Maternal impression of educational materials | Postpartum (<= 6 weeks)
  Mothers will be administered a brief survey (Likert scale) regarding how useful the respective book or brochure were to help them understand safe sleep practices and the importance of infant reading. They will also be asked if they still have the materials and how often they have reviewed them at home.
Clinical provider impression of educational materials | Prenatal/baseline visit (>=32 weeks gestation)
  Obstetric attending and resident physicians will be administered a brief survey (Likert scale) after the prenatal visit regarding how useful the respective book or brochure was to catalyze discussion of safe sleep and infant reading with the mother, with emphasis on feasibility in clinical practice.

SECONDARY OUTCOMES:
Home Literacy Orientation | Baseline prenatal (>= 32 weeks) and postpartum (<= 6 weeks).
  Prenatally, the mother will be administered a brief survey regarding the age at which the mother plans to begin reading with her infant (open-ended), planned frequency of reading (days per week), estimated number of children's books in the home, impression of the usefulness of reading to infants before 2 months old, and the value of discussing reading during prenatal visits (Likert scales). At the postpartum visit, this survey will be expanded to involve access to books, actual reading frequency, home reading routines, and the child's interest in being read to. An additional item regarding attitudes towards reading at home adapted from published research ("What are your 3 favorite things to do with your child these days?", noting if reading is mentioned) will also be asked.
DialogPR-I/T | Postpartum (<= 6 weeks).
  This is an 10-item parental report assessment of shared reading quality created by the principal investigator for caregivers of children under 18 months, based on a conceptual model of practices thought to enhance the reading experience and benefit child development. Score is 0-30 points, with higher score suggesting more nurturing reading behaviors.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Available in a de-identified fashion by written request & approval.

REFERENCES:
- [Background] Hutton JS, Gupta R, Gruber R, Berndsen J, DeWitt T, Ollberding NJ, Van Ginkel JB, Ammerman RT. Randomized Trial of a Children's Book Versus Brochures for Safe Sleep Knowledge and Adherence in a High-Risk Population. Acad Pediatr. 2017 Nov-Dec;17(8):879-886. doi: 10.1016/j.acap.2017.04.018. Epub 2017 Apr 24. PMID 28450082
- [Background] Hutton JS, Lin L, Gruber R, Berndsen J, DeWitt T, Van Ginkel JB, Ammerman RT. Shared Reading and Television Across the Perinatal Period in Low-SES Households. Clin Pediatr (Phila). 2018 Jul;57(8):904-912. doi: 10.1177/0009922817737077. Epub 2017 Oct 25. PMID 29067842
- [Derived] Hutton JS, Huang G, Crosh C, DeWitt T, Ittenbach RF. Shared reading with infants: SharePR a novel measure of shared reading quality. Pediatr Res. 2023 Mar;93(4):976-984. doi: 10.1038/s41390-022-02178-6. Epub 2022 Jul 19. PMID 35854086